CLINICAL TRIAL: NCT06693622
Title: Patient Preferences for Barrett's Esophagus and Esophageal Cancer Screening Tests: A Discrete Choice-Based Conjoint Analysis
Brief Title: Patient Preferences for Barrett's Esophagus and Esophageal Cancer Screening Tests
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other); University of California, Los Angeles (Other); University of Michigan (Other); Exact Sciences Corporation (Industry); VA Medical Center-West Los Angeles (U.S. Federal Agency); University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23-1758
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Gastro Esophageal Reflux Disease; Barrett Esophagus
Keywords: Gastroesophageal Reflux Disease; Barrett's Esophagus; Barrett's Esophagus Screening; BE; GERD
MeSH Terms: conditions — Gastroesophageal Reflux; Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: 556 eligible patients will be recruited across 5 participating sites to complete a discrete choice-based conjoint survey. The survey will be distributed to eligible patients via Sawtooth internet survey at the time of a clinic appointment or remotely via video chat.
  Interventions: Behavioral: Patient survey

INTERVENTIONS:
Behavioral: Patient survey — To assess patient preferences and barriers for attributes of BE/EAC screening modalities patients will complete a survey evaluating 5 domains: benefit of detection (sensitivity), convenience (time, setting), screening related physical harms (procedural discomfort), and financial harms. Prior to distribution, the survey will be refined and pretested among a sample of 5 patients.

SUMMARY:
This study plans to learn more about what patients think about screening for esophageal cancer (EAC) and Barrett's esophagus (BE); a pre-cancerous condition associated with esophageal cancer. The plan is to use this information to modify screening practices in the United States with the goal to decrease the number of people who die from esophageal cancer.

DETAILED DESCRIPTION:
To achieve this goal, patient preferences for BE/EAC screening tests will be evaluated through a prospective multicenter discrete choice-based conjoint survey. Patients will choose between a series of hypothetical options and rank their priorities and what they value according to differences in benefit of detection (sensitivity), convenience (time, setting), screening related physical harms (procedural discomfort), and financial harms. By evaluating relative importance of test characteristics and patient prioritization the study will (1) define patient preferences and barriers for attributes of BE/EAC screening modalities to elicit the overall preferred test as well as differences in each attribute that informed that choice and (2) characterize differences in BE/EAC test preferences by patient sociodemographic characteristics (age, sex, race, ethnicity) and by the presence or absence of gastroesophageal reflux disease (GERD).

ELIGIBILITY:
Inclusion Criteria:

* Provision to sign and date the consent form.
* Stated willingness to comply with all study procedures and be available for the duration of the study.
* Individual has 3 or more established risk factors for BE (age > 50 years, chronic GERD, male, white race, smoking, obesity, family history of BE/EAC).

Exclusion Criteria:

* Unable to consent.
* Prior diagnosis of BE/EAC.
* Life limiting comorbidity/ disability.
* Active dementia/ cognitive impairment.
* Incarcerated.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with 3 or more established risk factors for BE who have at least one outpatient clinic visit at a participating site. Patients will be identified at primary care and family medicine clinics. Patients with prior diagnosis of BE/EAC will be excluded. Across the 5 sites, planned enrollment is 556.
Sampling Method: Non-Probability Sample
Enrollment: 556 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Define patient preferred BE/EAC screening test and barriers for attributes of BE/EAC screening tests | Baseline
  A discrete choice-based conjoint analysis survey evaluating 5 domains: benefit of detection (sensitivity), convenience (time, setting), screening related physical harms (procedural discomfort), and financial harms will be used to determine the relative importance of BE/EAC screening test characteristics and patient priorities. Survey data will be reported in aggregate and factors and choices will be analyzed using the Fisher Exact and Mann-Whitney rank-sum tests. This approach will elicit the overall preferred test and differences in each test attribute that informed the patients choice.

SECONDARY OUTCOMES:
Characterization of differences in BE/EAC test preferences by patient sociodemographic characteristics and by patient presence or absence of GERD | Baseline
  Using the discrete choice-based conjoint analysis survey analysis, a logistic regression model of patient-specific attributes (age, sex, race, ethnicity) and by presence or absence of GERD will be used to evaluate if disparities in patient demographics or heath history impact complex decision making.

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Wani, MD, Principal Investigator — University of Colorado, Denver; Jennifer Kolb, MD, MS, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in original publications after deidentification (text, tables, figures, appendixes).
Supporting Information: Study Protocol
Time Frame: 9 months to 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal and investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  These data can only be used for individual participant data meta-analysis.